CLINICAL TRIAL: NCT04899947
Title: Children, Adolescents and Their Providers: the Narcolepsy Assessment Partnership (CATNAPTM)
Brief Title: Child and Adolescent Registry for Participants With Narcolepsy
Status: Recruiting | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: HealhieCATNAPN.A.
Record Dates: First submitted 2021-04-30; First posted 2021-05-25 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
CATNAP is a patient registry designed to improve the understanding of the natural history of narcolepsy in pediatric patients. Descriptive statistics on disease characteristics will be performed.

The study has 16 active clinical sites and a virtual site that widens participation to anywhere in the United States. For more information about the study or to access the Online Patient Enrollment System, visit the CATNAP website: https://catnap.healthie.net/welcome or email catnap@pulseinfoframe.com. The Online Patient Enrollment System, CATNAP website, can also be found in the references section.

ELIGIBILITY:
Inclusion Criteria:

* Any child or adolescent with a physician-confirmed diagnosis of narcolepsy
* Age less than 18 years
* Willing to participate in the Registry and complete the informed consent form
* Able to participate in English based registry

Exclusion Criteria:

* Age 18 years or more
* Fail to complete the informed consent form

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child or adolescent with a physician-confirmed diagnosis of narcolepsy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Improve Understanding of Natural History of Pediatric Narcolepsy | Up to 4 years
Characterize the Presentation, Identification, and Diagnosis of Narcolepsy in Pediatric Participants | Up to 4 years
Understand Treatment Practices and Outcomes Captured by Treatment Regimen and Rational for Changes | Up to 4 years

SECONDARY OUTCOMES:
Improvements in Quality of Life (QoL) as Measured by Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) Questionnaire | Up to 4 years
QoL - Pediatric Quality of Life Inventory (PedsQL) | Up to 4 years
Change in frequency of child ehavioral problems utilizing the Child Behavior Checklist (CBCL) | Up to 4 years
Patient Reported Outcomes Measurement Information System (PROMIS) Peer Relationship-Parent Proxy Short Form v2.0 | Up to 4 years
Caregiver Work Limitations Questionnaire (C-WLQ) | Up to 4 years
Work Productivity and Activity Impairment (WPAI) | Up to 4 years
Change in Caregiver Well-being Measured by the Caregiver Well-Being Scale (Shortened) | Up to 4 years
Change in Level of Social Support using the Social Support Survey Instrument | Up to 4 years
Change in Pittsburgh Sleep Quality index (PSQI) scores | Up to 4 years

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of Arkansas, Fayetteville, Arkansas
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Stanford University, Redwood City, California
  - University of California San Diego, San Diego, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Research Institute, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Trinity Health-Michigan, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Michigan
  - St. Luke's Hospital, Chesterfield, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Northwell Health, Manhasset, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Centre (UHCMC), Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Geisinger, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - Children's Hospital of the King's Daughters, Norfolk, Virginia

REFERENCES:
- See also: Online Patient Enrollment System — https://catnap.healthie.net/welcome